CLINICAL TRIAL: NCT04603131
Title: Phase-I Open Label, Dose-escalation Clinical Trial to Evaluate the Safety, Tolerability and Immunogenicity of Chikungunya Vaccine in Healthy Adults of 18 to 50 Years Age
Brief Title: Clinical Trial to Evaluate the Immunogenicity of Chikungunya Vaccine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bharat Biotech International Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: BBIL/CHIKV/I/2014
Record Dates: First submitted 2017-07-17; First posted 2020-10-26 (Actual); Last update posted 2020-10-28 (Actual); Status verified 2020-10

CONDITIONS: Chikungunya
MeSH Terms: conditions — Chikungunya Fever

STUDY DESIGN:
Intervention Model Description: Chikungunya vaccine is an inactivated virus vaccine. There will be three study arms and subjects will be vaccinated in a dose escalation manner.In each arm, vaccine will be administered on day1, day29, day57. Vaccine will be administered through intramuscular route.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- BBV87 - 10 mcg (Experimental): Inactivated Chikungunya virus vaccine (BBV87) in three dose strengths (10, 20 and 30 mcg) administered intramuscularly on Day 0, 29 and 57
  Interventions: Biological: Inactivated Chikungunya virus vaccine 10 mcg
- Placebo (Placebo Comparator): Placebo administered intramuscularly on Day 0, 29 and 57
  Interventions: Biological: Placebo
- BBV87 -30 mcg (Experimental): Inactivated Chikungunya virus vaccine (BBV87) in three dose strengths administered intramuscularly on Day 0, 29 and 57
  Interventions: Biological: Inactivated Chikungunya virus vaccine 20 mcg
- BBV87 -20 mcg (Experimental): Inactivated Chikungunya virus vaccine (BBV87) in three dose strengths administered intramuscularly on Day 0, 29 and 57
  Interventions: Biological: Inactivated Chikungunya virus vaccine 30 mcg

INTERVENTIONS:
Biological: Inactivated Chikungunya virus vaccine 20 mcg — 3 doses of Inactivated Chikungunya virus vaccine (BBV87) administered intramuscularly on Day 0, 29 and 57
  Arms: BBV87 -30 mcg
Biological: Inactivated Chikungunya virus vaccine 30 mcg — 3 doses of Inactivated Chikungunya virus vaccine (BBV87) administered intramuscularly on Day 0, 29 and 57
  Arms: BBV87 -20 mcg
Biological: Inactivated Chikungunya virus vaccine 10 mcg — 3 doses of Inactivated Chikungunya virus vaccine (BBV87) administered intramuscularly on Day 0, 29 and 57
  Arms: BBV87 - 10 mcg
Biological: Placebo — 3 doses of Placebo administered intramuscularly on Day 0, 29 and 57
  Arms: Placebo

SUMMARY:
Chikungunya vaccine is an inactivated virus vaccine. There will be three study arms and subjects will be vaccinated in a dose escalation manner.In each arm, vaccine will be administered on Day 1, Day 29, and Day 57. Vaccine will be administered through intramuscular route.

DETAILED DESCRIPTION:
This is an open label phase I study for assessing the safety, tolerance and immunogenicity of 3 escalated doses of the test vaccine, BBV87. The study design has four treatment groups - 3 test groups and a control placebo group with 15 subjects in each group. However, the groups will be divided into three study arms: each arm will have 15 subjects of the test vaccine group and 5 subjects of the placebo group. The randomization will be done in a way that allots 5 subjects of the placebo group to each test dose group. All subjects will be screened (via medical history, physical examination and laboratory investigations) to establish the eligibility criteria. This includes negative antibodies, CHIKV IgG, by ELISA method. The test vaccine and placebo will be administered as 3 doses at 28 days interval on day 1±2, 29±2, and 57±2. Vaccine administration will be performed as an in-patient procedure. Subjects will be admitted in CPU 24 hrs prior to vaccine administration, and will be shifted to MICU for vaccination and observed for 48 hrs; and will be discharged upon completion of all clinical monitoring procedures. Laboratory and biochemical tests will be performed as part of clinical monitoring before discharge, and 24 hrs after vaccine administration. Following vaccination, all participants will be monitored throughout the study period for adverse events with daily telephone contacts (for 7 days after each vaccine, and then weekly), interim clinic visits, subject diary cards, and haematological & biochemical laboratory tests.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 and ≤50 yrs inclusive on the day of screening
* Able and willing to complete informed consent process with understanding of the purpose and procedures of the study
* Medical history and physical examination without clinically significant findings at the time of screening
* Haematological and biochemical values either within institutional normal range and accompanied by physician approval
* Agree to keep a daily record of symptoms for the duration of the study
* Available for clinical follow-up throughout the study period via telephone contact as well as clinic visits

Female specific criteria:

* If female of child bearing potential- have a negative urine pregnancy test result within 24 hrs of the scheduled first vaccination

Exclusion Criteria:

Female specific criteria:

* Woman who is breast feeding or planning to become pregnant during the study period.

General Criteria:

* History of suspected or confirmed Chikungunya fever

(Case definition for Suspected Chikungunya: A subject meeting both the clinical and epidemiological criteria.

* Clinical criteria: acute onset of fever >38.5°C and severe arthralgia/arthritis not explained by other medical conditions.
* Epidemiological criteria: residing or having visited epidemic areas, having reported transmission within 15 days prior to the onset of symptoms.

Case definition for Confirmed Chikungunya:

A subject meeting the laboratory criteria of positive ELISA test for CHIKV IgG.)

* Clinically significant abnormal clinical laboratory values including blood pressure(>140 mmHg systolic and >90 mmHg diastolic) when 3 measurements are taken 30 min apart , in seating position and at rest
* Body mass index (BMI) ≥ 25 [BMI will be calculated as weight in Kilograms/(height in metres)2]
* Test positive for HIV or Hepatitis B infection
* History of cardiovascular disease
* History of immune deficiency or autoimmune disease
* Have active or history of arthritis (joint swelling, pain, tenderness, warmth or erythema) within the last 6 months from date of screening
* Have an active or history of malignant conditions including haematological malignancy
* Have a history of degenerative neurological disease (e.g. GuillainBarre Syndrome, multiple sclerosis)
* Have received any vaccination within 4 weeks prior to the vaccination in this study
* Have received blood transfusion or immunoglobulin within 30 days prior to vaccination in this study
* Have a history of serious reactions to any vaccines that preclude receipt of study vaccinations as determined by the investigator
* Have asthma that is unstable or required emergent care, urgent care, hospitalization or intubation during the past two years or that is expected to require the use of oral or intravenous corticosteroids
* Have diabetes mellitus (type I or II), with the exception of history of gestational diabetes
* Have received any investigational drug in 6 weeks prior to screening
* Is currently participating in any form of clinical trial that involves intervention.
* Is likely to participate in any other clinical trial during the study period.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2017-04-17 (Actual); Primary Completion 2018-01-30 (Actual); Study Completion 2018-07-30 (Actual)

PRIMARY OUTCOMES:
Occurrence of adverse events and Serious Adverse events post each dose | Within 24 hrs
  safety
Occurrence of adverse events and Serious Adverse events post each dose | 7 Days,
  safety
Occurrence of adverse events and Serious Adverse event 28 days after the last dose of vaccine | 9 months
  safety

SECONDARY OUTCOMES:
Immunogenicity in terms of GMT estimated by 50 percent plaque reduction neutralization test | day 28
  Immunogenicity
Immunogenicity in terms of GMT estimated by 50 percent plaque reduction neutralization test | day 56
  Immunogenicity
Immunogenicity in terms of GMT estimated by 50 percent plaque reduction neutralization test | day 84
  Immunogenicity
Proportion of subjects with four fold seroconversion | day 28
  Immunogenicity
Proportion of subjects with four fold seroconversion | day 56
  Immunogenicity
Proportion of subjects with four fold seroconversion | day 84
  Immunogenicity

CONTACTS AND LOCATIONS:
Overall Officials: Krishna Mohan, PHD, Study Director — Bharat Biotech International Limited
Locations (4):
- India (4):
  - King George Hospital, Visakhapatnam, Andhra Pradesh
  - Medanta - The Medicity, Gurgaon, Haryana
  - KEM Hospital, Mumbai, Maharashtra
  - Panchsheel Hospital, Delhi

IPD SHARING:
Plan to Share IPD: No